CLINICAL TRIAL: NCT03960086
Title: Effectiveness of Custom-made Foot Orthoses vs Heel Lifts in Children With Calcaneal Apophysitis (Sever Disease): a Randomized Controlled Trial
Brief Title: Effectiveness of Custom-made Foot Orthoses vs Heel Lifts in Children With Calcaneal Apophysitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Podoactiva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sever insoles-heel lifts
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Calcaneal Apophysitis; Sever's Disease

STUDY DESIGN:
Intervention Model Description: The study was a parallel-group, randomized controlled trial with concealed allocation, blinding of investigators and assessors and intention-to-treat analysis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made foot orthoses (Experimental): Children in the experimental group received as treatment intervention custom-made polypropylene foot orthoses (Podoactiva®, Spain). They were advised pragmatically to wear the orthoses at least 8 to 10 hours per day for the daily life and during sport activity.
  Treatment period of 12 weeks
  Interventions: Other: Podoactiva cutom-made foot orthoses
- Heel Lifts (Active Comparator): Children in the experimental group received as treatment intervention custom-made polypropylene foot orthoses (Podoactiva®, Spain). They were advised pragmatically to wear the orthoses at least 8 to 10 hours per day for the daily life and during sport activity.
  Treatment period of 12 weeks
  Interventions: Other: Podoactiva heel lifts

INTERVENTIONS:
Other: Podoactiva cutom-made foot orthoses — Children had to use the orthotics daily during the intervention period
  Arms: Custom-made foot orthoses
Other: Podoactiva heel lifts — Children had to use the orthotics daily during the intervention period
  Arms: Heel Lifts

SUMMARY:
The study was a parallel-group, randomized controlled trial with concealed allocation, blinding of investigators and assessors and intention-to-treat analysis. It examined the effect of custom-made foot orthoses and heel lifts in children with calcaneal apophysitis.

It was hypothesized that the primary outcome, pain relief, would be significantly improved with the custom-made orthosis compared to the heel lift.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed radiologically with calcaneal osteochondritis
* diagnosed radiologically with calcaneal osteochondritis
* have signed informed consent

Exclusion Criteria:

* had suffered some trauma on the heel in the past 2 months
* had received anti-inflammatory drugs and/or physical treatment for pain in the past 3 months
* had presented physical or neurological impairment
* were not interested

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Visual analogical scale (VAS) | At baseine and after the intervention period
  Subjective Sever´s disease pain perception before and after the intervention measured by the Visual analogical scale (VAS)
Algometry | At baseine and after the intervention period
  Pressure-pain threshold measured in the heel in Sever´s disease, before and after the intervention
Sport activity pain perception | At baseine and after the intervention period
  Sever´s disease pain perception measured asking the following question: "Do you have pain at sport activity?", before and after intervention

SECONDARY OUTCOMES:
Foot Posture Index (FPI) | At baseline
  values of Foot Posture Index (FPI) test in children with calcaneal apophysistis
lunge test values | At baseline
  values of lunge test in children with calcaneal apophysistis

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandro Jesús Almenar Arasanz, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
No, participants in this study were not adults and in the informed consent signed there was not indiated this statment

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03960086/Prot_SAP_000.pdf